CLINICAL TRIAL: NCT06572670
Title: The Effect of Progressive Relaxation Exercise Performed Before Coronary Angiography on Anxiety, Comfort, Pain and Physiological Parameters
Brief Title: The Effect of Progressive Relaxation Exercise Performed Before Coronary Angiography
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Sevda Korkut, Associate Prof., TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024/30
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Coronary Angiography; Progressive Relaxation Exercise; Nursing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive relaxation exercise before coronary angiography (Experimental): Patients in the intervention group will undergo progressive relaxation before undergoing angiography.
  Interventions: Other: Progressive relaxation exercise before coronary angiography
- Control group (No Intervention): No application will be made to the control group before the procedure.

INTERVENTIONS:
Other: Progressive relaxation exercise before coronary angiography — Patients in the intervention group will undergo progressive relaxation before undergoing angiography.
  Arms: Progressive relaxation exercise before coronary angiography

SUMMARY:
This study was planned to examine the effects of progressive relaxation exercise on anxiety, comfort, pain and physiological parameters in patients undergoing coronary angiography. The data of the study will be collected using the Descriptive Characteristics Questionnaire Form, State and Trait Anxiety Inventory, Perianesthesia Comfort Questionnaire, Visual Analog Scale (VAS), Vital Signs Follow-up Form, Complication Follow-up Form and Progressive Relaxation Exercise Application Guidelines.

DETAILED DESCRIPTION:
This study was planned to examine the effects of progressive relaxation exercise on anxiety, comfort, pain and physiological parameters in patients undergoing coronary angiography. The data of the study will be collected using the Descriptive Characteristics Questionnaire Form, State and Trait Anxiety Inventory, Perianesthesia Comfort Questionnaire, Visual Analog Scale (VAS), Vital Signs Follow-up Form, Complication Follow-up Form and Progressive Relaxation Exercise Application Guidelines. Patients in the intervention group will undergo progressive relaxation before undergoing angiography. Standard practices of the clinic will be applied to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients who can speak and understand Turkish,
* Are over 18 years old,
* Have space and time orientation,
* Will undergo coronary angiography for the first time,
* Do not have any psychiatric illness,
* Do not have vision or hearing problems,
* Volunteer to participate in the study will be included.

Exclusion Criteria:

* Patients who experience any pain or have chronic pain before coronary angiography,
* Patients who use antihistamines and psychiatric medications,
* Patients who do not volunteer to participate in the study,
* Patients who have undergone orthopedic surgery or have any medically diagnosed health problems (orthopedic, neurological, psychological) that prevent relaxation exercises,
* Patients who have taken sedatives or painkillers up to 5 hours before coronary angiography will not be included in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Anxiety level | 30 minutes after angiography
  This inventory, which consists of a total of 40 items, is analyzed in two separate sections: The first part is the State Anxiety Inventory, which consists of 20 items, and the individual answers this section with his/her current feelings. The second part is the Trait Anxiety Inventory, which also consists of 20 items, and the individual answers this section with the feelings they have felt in the last 7 days.
Comfort level | 30 minutes after angiography
  The scale, which is based on the concept of comfort, consists of a total of 24 items, 12 of which question the comfort status of the individual before and after the surgical intervention, 12 of which question positive and 12 of which question negative experiences.
Pain level | 30 minutes after angiography
  Pain will be assessed with the Visual Analog Scale. This scale consists of a 10 cm line with values between 0 and 10. The beginning of the line (number 0) indicates "no pain", while the end of the line (number 10) indicates the most severe pain.

SECONDARY OUTCOMES:
Blood pressure to be assessed with monitor | 30 minutes after angiography
  The patient's blood pressure will be measured from the brachial artery with a bedside monitor and the result will be recorded in mmHg.
Pulse to be assessed with monitor | 30 minutes after angiography
  Heart rate will be measured with a bedside monitor that can be measured from a finger and recorded as beats/min.
Respiratory rate | 30 minutes after angiography
  Respiratory rate will be measured by counting the number of inspirations and expiration from the patient's chest movements.

IPD SHARING:
Plan to Share IPD: No